CLINICAL TRIAL: NCT04078516
Title: Perception Threshold Tracking(PTT): A Novel Method for Early Detection and Grading of Diabetic Peripheral Neuropathy
Brief Title: Methods of Early Detection and Grading Of Diabetic Peripheral Neuropathy (MEDON)
Acronym: MEDON
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Niels Ejskjær, Professor of Endocrinology, Aalborg University Hospital
Other Study IDs: N-20190003
Record Dates: First submitted 2019-08-28; First posted 2019-09-06 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Neuropathy, Diabetic; Neuropathy, Painful
Keywords: diabetes; neuropathy; early detection; small nerve fibers
MeSH Terms: conditions — Diabetic Neuropathies; Neuropathy, Painful; Diabetes Mellitus | interventions — Laser-Doppler Flowmetry; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Type 1 diabetes and painful neuropathy: No interventions. A series of observationel/expirimental methods for detecting and grading neuropathy will be applied.
  Interventions: Diagnostic Test: Perception Threshold Tracking (PTT); Diagnostic Test: Axon-flair mediated respons; Diagnostic Test: Heart rate variability; Diagnostic Test: Quantitative Sensory Testing (QST); Diagnostic Test: Peripheral blood pressure and transcutaneous oxygen tension; Diagnostic Test: Magnetic Resonance Imaging (MRI); Diagnostic Test: Questionnaires; Diagnostic Test: Corneal Confocal Microscopy /CCM)
- Type 1 diabetes and non-painful neuropathy: No interventions. A series of observationel/expirimental methods for detecting and grading neuropathy will be applied.
  Interventions: Diagnostic Test: Perception Threshold Tracking (PTT); Diagnostic Test: Axon-flair mediated respons; Diagnostic Test: Heart rate variability; Diagnostic Test: Quantitative Sensory Testing (QST); Diagnostic Test: Peripheral blood pressure and transcutaneous oxygen tension; Diagnostic Test: Magnetic Resonance Imaging (MRI); Diagnostic Test: Questionnaires; Diagnostic Test: Corneal Confocal Microscopy /CCM)
- Type 1 diabetes and no neuropathy: No interventions. A series of observationel/expirimental methods for detecting and grading neuropathy will be applied.
  Interventions: Diagnostic Test: Perception Threshold Tracking (PTT); Diagnostic Test: Axon-flair mediated respons; Diagnostic Test: Heart rate variability; Diagnostic Test: Quantitative Sensory Testing (QST); Diagnostic Test: Peripheral blood pressure and transcutaneous oxygen tension; Diagnostic Test: Magnetic Resonance Imaging (MRI); Diagnostic Test: Questionnaires; Diagnostic Test: Corneal Confocal Microscopy /CCM)
- Matched controls without diabetes: No interventions. A series of observationel/expirimental methods for detecting and grading neuropathy will be applied.
  Interventions: Diagnostic Test: Perception Threshold Tracking (PTT); Diagnostic Test: Axon-flair mediated respons; Diagnostic Test: Heart rate variability; Diagnostic Test: Quantitative Sensory Testing (QST); Diagnostic Test: Peripheral blood pressure and transcutaneous oxygen tension; Diagnostic Test: Magnetic Resonance Imaging (MRI); Diagnostic Test: Questionnaires; Diagnostic Test: Corneal Confocal Microscopy /CCM)

INTERVENTIONS:
Diagnostic Test: Perception Threshold Tracking (PTT) — low-current electrical stimulation of both large- and small nerve fibers.
Diagnostic Test: Axon-flair mediated respons — Laser-doppler examination of small blood vessels in the peripheral skin.
  Other Names: Laser-doppler
Diagnostic Test: Heart rate variability — 4 measurements of heart rate.
  Other Names: Vagus TM
Diagnostic Test: Quantitative Sensory Testing (QST) — Seven tests measuring 13 parameters including heat- and cold-detection and pain thresholds, mechanical pain treshold, mechanical detection threshold, pressure pain treshold and vibration threshold.
  Other Names: German Research Network on Neuropathic Pain (DFNS) standard protocol
Diagnostic Test: Peripheral blood pressure and transcutaneous oxygen tension — Ankle/brachial index, toe/brachial index, TcpO2.
  Other Names: Perimed 6000
Diagnostic Test: Magnetic Resonance Imaging (MRI) — MRI-scans of peripheral nerves and the central nervous system. Blood oxygen level dependent (BOLD) MRI.
Diagnostic Test: Questionnaires — Questionnaires for detecting painful neuropathy
  Other Names: PainDETECT, Douleur Neuropathique 4
Diagnostic Test: Corneal Confocal Microscopy /CCM) — Confocal microscopy of the cornea measuring NBD, NFD, NFL

SUMMARY:
MEDON aims to examine new methods for early detection and grading of diabetic peripheral neuropathy focusing on both small- and large nerve fibers. Furthermore, MEDON aims to describe differences between people with classic diabetic peripheral neuropathy and those with painful diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women minimum 18 years of age and maximum 75 years of age
2. Signed informed consent form
3. Diagnosed with diabetes type I (for group 1-3)
4. Diagnosed with DPN defined as a threshold above 25-volt biothesiometry or absent feeling on the big toe using 10g-monofilament. (for group 1-2)
5. Answered questionnaire: PainDETECT
6. Nothing abnormal on initial tests (group 4)
7. Accepted initial screening blood samples
8. MRI-compatible participant

Exclusion Criteria:

* 1. Current or previous alcohol- or drug abuse 2. Abnormal screening blood samples 3. Not being able to understand Danish written and/or verbally 4. Not being able to corporate to examination (e.g. not being able to speak, suffering from senile dementia etc.) 5. Previous chemotherapy or intake of experimental medicine 6. Active HSV- or VZV-infection or known HIV 7. Known severe skin disease 8. Known neural damage or disease in the neural system (e.g. MS, Guillain-Barre etc.) 9. Critical limb ischemia defined as in current clinical consensus 10. Allergy or intolerance to histamine or inability to make do without for one day 11. Pregnancy 12. Active cancer-disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population include four well-defined groups of subjects:
  1. Patients with Type 1 diabetes and painful diabetic peripheral neuropathy (DPN).
  2. Patients with Type 1 diabetes and non-painful diabetic peripheral neuropathy (DPN)
  3. Patients with Type 1 diabetes and without diabetic peripheral neuropathy (VPT<15) (DPN).
  4. Healthy control subjects matched for age, BMI, and gender. Diabetes duration, HbA1c, insulin use, ethnicity, and co-morbidities will be matched between group 1, 2 and 3 to best ability.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic value of CCM, PTT, AF and MRI | End of study (when all patients have completed all sessions. Latest 31. december 2021)
  Using Quantitative Sensory Testing (small fibers) and conventional nerve conduction studies (large fibers) as golden standards, we will determine the prognostic value of:
  Perception Threshold Tracking Corneal Confocal Microscopy Axon-flair mediated response MRI-scans in detecting neuropathy. Sensitivity and specificity will be reported.
  OBS! Tests will be tested in the initial groups and AFTER a group re-arrangement based on results from QST and NCS.

SECONDARY OUTCOMES:
Validation of PainDETECT in diabetes | End of study / end of inclusion (when all patients have completed the screening session. Latest 31. november 2021)
  Correlation between PainDETECT and DN4 will be reported.

OTHER OUTCOMES:
Exploratory measures | End of study (latest december 31 2021).
  An multi-variant analysis to determine the predictive ability of combinations of primary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Ejskjær, Professor, Principal Investigator — Steno Diabtes Center North Denmark, Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with collaborating department: Department of Radiology with the purpose of analyzing the data and comparing it to their MRI scans.
  Data will be shared with Aalborg University with the purpose of analyzing data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: During and after the study. Data will be available no longer than needed for analyzing.
Access Criteria: anonymized data

REFERENCES:
- [Derived] Moussa F, Taleb S, Borbjerg MK, Croosu SS, Morch CD, Frokjaer JB, Hansen TM, Ejskjaer N, Roikjer J. Corneal Immune Cells and Their Relation to Diabetic Peripheral Neuropathy and Neuropathic Pain. Muscle Nerve. 2026 Jan;73(1):72-78. doi: 10.1002/mus.70061. Epub 2025 Nov 17. PMID 41246983
- [Derived] Roikjer J, Croosu SS, Sejergaard BF, Hansen TM, Frokjaer JB, Sondergaard CB, Petropoulos IN, Malik RA, Nielsen E, Morch CD, Ejskjaer N. Diagnostic Accuracy of Perception Threshold Tracking in the Detection of Small Fiber Damage in Type 1 Diabetes. J Diabetes Sci Technol. 2024 Sep;18(5):1157-1164. doi: 10.1177/19322968231157431. Epub 2023 Feb 24. PMID 36825610
- [Derived] Roikjer J, Croosu SS, Frokjaer JB, Hansen TM, Arendt-Nielsen L, Ejskjaer N, Morch CD. Perception threshold tracking: validating a novel method for assessing function of large and small sensory nerve fibers in diabetic peripheral neuropathy with and without pain. Pain. 2023 Apr 1;164(4):886-894. doi: 10.1097/j.pain.0000000000002780. Epub 2022 Sep 19. PMID 36130086

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT04078516/Prot_SAP_000.pdf